CLINICAL TRIAL: NCT06747091
Title: Adjuvant Ablation for PeRsistent AtrIal FibrillAtion Using Dual ENergy LatticE Tip Catheter: ARIADNE-Randomized Clinical Trial
Brief Title: ARIADNE Clinical Trial
Acronym: ARIADNE RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stavros E Mountantonakis (Other)
Responsible Party: Sponsor-Investigator, Stavros E Mountantonakis, Director, Cardiac Electrophysiology, Northwell Health
Organization: Northwell Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-0935-LHH
Record Dates: First submitted 2024-11-04; First posted 2024-12-24 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Pulsed Field Ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to the ablation strategy they are randomized to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PVI using PFA energy (Active Comparator): Pulmonary vein isolation using PFA energy
  Interventions: Procedure: Catheter Ablation
- PVI and posterior wall isolation using PFA energy (Active Comparator): Pulmonary vein isolation and posterior wall isolation using PFA energy
  Interventions: Procedure: Catheter Ablation
- PVI and posterior wall isolation (PFA) and mitral isthmus ablation using RFA or PFA energy. (Active Comparator): Pulmonary vein isolation and posterior wall isolation (PFA) and mitral isthmus ablation using RFA or PFA energy.
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — This is a prospective randomized clinical trial. Patients will undergo catheter ablation for persistent AF using a lattice-tip catheter that can switch between RFA and PFA energy. Enrolled patients will be randomized to one of three ablation strategies:

SUMMARY:
A prospective multi-arm parallel group randomized clinical trial to compare the efficacy of three ablation strategies in patients with persistent atrial fibrillation using using a lattice-tip catheter that can switch between RFA and PFA energy. The incremental benefit of posterior wall isolation (PWI) and mitral isthmus ablation may contribute to greater freedom from atrial fibrillation at twelve months.

DETAILED DESCRIPTION:
This is a prospective randomized clinical trial. Patients will undergo catheter ablation for persistent AF using a lattice-tip catheter that can switch between RFA and PFA energy. Enrolled patients will be randomized to one of three ablation strategies:

1. Pulmonary vein isolation using PFA energy
2. Pulmonary vein isolation and posterior wall isolation using PFA energy
3. Pulmonary vein isolation and posterior wall isolation (PFA) and mitral isthmus ablation using RFA or PFA energy.

Patients will receive an implantable loop recorder prior to, during or post index ablation procedure for continuous monitoring for clinical recurrence of AF/AT/AFL

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic PerAF documented by

(1a) a physician's note indicating symptoms consistent with AF sustained longer than 7 days but less than 12 months; AND electrocardiographic evidence

2. . Suitable candidate for catheter ablation.

3. . Adults aged 18 - 80 years.

4. . Willing and able to comply with all baseline and follow-up evaluations for the full length of the study.

Exclusion Criteria:

1. AF secondary to electrolyte imbalance, thyroid disease, acute alcohol intoxication, or other reversible or non-cardiac cause.
2. Previous left atrial ablation or surgical procedure (including septal closure or left atrial appendage closure).
3. Valvular cardiac surgical/percutaneous procedure (e.g., ventriculotomy, atriotomy, and valve repair or replacement and presence of a prosthetic valve).
4. Any carotid stenting or endarterectomy.
5. Any cardiac procedure (surgical or percutaneous) or percutaneous coronary intervention within the 90 days prior to the initial procedure.
6. Coronary artery bypass graft (CABG) procedure within the 6 months prior to the initial procedure.
7. Awaiting cardiac transplantation or other cardiac surgery within the 12 months following the initial ablation procedure.
8. Documented thromboembolic event (stroke or transient ischemic attack) within 6 months (180 days) prior to the initial ablation procedure.
9. Documented left atrial thrombus on imaging.
10. History of blood clotting or bleeding abnormalities.
11. Any condition contraindicating chronic anticoagulation.
12. Myocardial infarction (MI) within the 3 months (90 days) prior to the initial procedure.
13. Body mass index >40 kg/m2.
14. Left atrial diameter >55 mm (anterioposterior).
15. Diagnosed atrial myxoma.
16. Uncontrolled heart failure or NYHA Class III or IV heart failure.
17. Rheumatic heart disease.
18. Hypertrophic cardiomyopathy.
19. Unstable angina.
20. Moderate to severe mitral valve stenosis.
21. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2).
22. Primary pulmonary hypertension.
23. Significant restrictive or obstructive pulmonary disease or chronic respiratory condition.
24. Renal failure requiring dialysis.
25. History of severe Gastroesophageal Reflux Disease (GERD) requiring surgical and/or mechanical intervention.
26. Acute illness, active systemic infection, or sepsis.
27. Contraindication to both computed tomography and magnetic resonance angiography.
28. Significant congenital anomaly or medical problem that, in the opinion of the investigator, would preclude enrollment in this study or compliance with follow-up requirements or would impact the scientific soundness of the clinical study results.
29. Current or anticipated participation in any other clinical study of a drug, device, or biologic during the duration of the study not pre-approved by the Sponsor.
30. Presence of intramural thrombus, tumor, or other abnormality that precludes vascular access, catheter introduction, or manipulation.
31. Known drug or alcohol dependency.
32. Life expectancy less than 12 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects free from primary effectiveness failure | 12 Months
  The primary effectiveness endpoint is freedom from documented recurrence of AF, atrial tachycardia (AT), or atrial flutter (AFL) lasting >2 minutes based on electrocardiographic data through 12-month follow-up and excluding a 60-day blanking period.

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Mountantonakis, MD, Principal Investigator — Northwell Health
Locations (3):
- United States (3):
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Kristie Coleman, New York, New York